CLINICAL TRIAL: NCT05881616
Title: Serum Metabolomics Analysis for Early Diagnosis and Pathogenesis of Gestational Diabetes Mellitus
Brief Title: Study on Serum Metabolomics of GDM
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Lu LI, Research Professor, Zhejiang University
Other Study IDs: IRB-20230193-R
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: GDM; Pathogenesis; Diagnosis
Keywords: Metabolomics
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GDM group: Pregnant women aged 20-40 with positive oral glucose tolerance test (OGTT) results at 24-28 weeks.
  Interventions: Other: Specimen samples and baseline data collection
- non-GDM group: Pregnant women aged 20-40 with negative OGTT results at 24-28 weeks.
  Interventions: Other: Specimen samples and baseline data collection
- Control group: Healthy non-pregnant women aged 20-40.
  Interventions: Other: Specimen samples and baseline data collection

INTERVENTIONS:
Other: Specimen samples and baseline data collection — The remaining serum samples from routine blood tests of subjects will be collected (without additional blood collection), with a serum sample size of approximately 1 mL per subject. The samples will be pre-processed and stored at ultra-low temperatures. At the same time, clinical baseline data of subjects will be collected from outpatient or inpatient medical records, including but not limited to age, height, weight, blood pressure, and gestational age.
  Groups: GDM group
Other: Specimen samples and baseline data collection — The remaining serum samples from routine blood tests of subjects will be collected (without additional blood collection), with a serum sample size of approximately 1 mL per subject. The samples will be pre-processed and stored at ultra-low temperatures. At the same time, clinical baseline data of subjects will be collected from outpatient or inpatient medical records, including but not limited to age, height, weight, blood pressure, and gestational age.
  Groups: non-GDM group
Other: Specimen samples and baseline data collection — The remaining serum samples from routine blood tests of subjects will be collected (without additional blood collection), with a serum sample size of approximately 1 mL per subject. The samples will be pre-processed and stored at ultra-low temperatures. At the same time, clinical baseline data of subjects will be collected from outpatient or inpatient medical records, including but not limited to age, height, weight, blood pressure, and gestational age.
  Groups: Control group

SUMMARY:
This study aims to collect serum samples from healthy non-pregnant women, pregnant women with and without Gestational Diabetes Mellitus (GDM). We will analyze the metabolite changes among the three groups using clinical metabolomics and identify potential biomarkers and metabolic pathways. This study will provide scientific evidence for early clinical diagnosis, prevention, control, and treatment research of GDM.

ELIGIBILITY:
Inclusion Criteria:

* No obvious abnormalities in all inspection items
* No history of diabetes
* No particular dietary habits
* No previous history of other mental illnesses
* No history of drug abuse or allergies
* No history of smoking or drinking

Exclusion Criteria:

* Pregnancy complications such as uterine fibroids, hyperthyroidism/hypothyroidism, and antiphospholipid antibody syndrome
* Critical illnesses such as cardiovascular disease or abnormal liver/kidney function
* Personal history of syphilis, HIV positive, and other infectious diseases
* Artificial insemination or IVF pregnancy
* Multiple pregnancy (twins or more)
* Patients participating in other clinical studies
* Other reasons that researchers think are inappropriate

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study aims to recruit pregnant women undergoing routine prenatal examinations and healthy women undergoing routine physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Content of serum metabolomics | Second trimester (24-28 gestational weeks)
  Based on non-targeted metabolomics technology, the metabolites in serum were comprehensively detected. Differential metabolites were screened using multivariate statistical analysis. Then quantitatively detect the content of these metabolites to find the differential metabolites with predictive ability for GDM.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Hangzhou, Zhejiang, China